CLINICAL TRIAL: NCT01049204
Title: Randomised, Placebo Controlled, Phase IV, Safety and Exploratory Immunogenicity Study on Maraviroc, an Oral ART CCR5 Inhibitor, on the Intensification of Immune Function in HIV-1 Infected Subjects Receiving Immunisation With Novel Antigens
Brief Title: Impact of Maraviroc on the Immune Function in HIV-1 Infected Subjects Receiving Immunisation With Novel Antigens
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The data from the first 48 patients recruited has now been analysed, and it has been determined that it is sufficient to meet the study objectives.
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSAT 030; EudraCT No. 2008-006769-95 (Other: EU Clinical Trials database)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: HIV Infections
Keywords: HIV; HIV-1 Infections
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): Nadir CD4 count >200 cells/µl blood and randomised to Maraviroc 150mg BD
  Interventions: Drug: Maraviroc
- Group 2 (Placebo Comparator): Nadir CD4 count >200 cells/µl blood and randomised to placebo twice daily for 24 weeks
  Interventions: Drug: placebo
- Group 3 (Active Comparator): Nadir CD4 count ≤200 cells/µl blood and randomised to Maraviroc 150mg BD
  Interventions: Drug: Maraviroc
- Group 4 (Placebo Comparator): Nadir CD4 count ≤200 cells/µl blood and randomised to placebo twice daily for 24 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 150 mg twice daily for 24 weeks
  Other Names: Celsentri
  Arms: Group 1; Group 3
Drug: placebo — Placebo twice daily for 24 weeks
  Arms: Group 2; Group 4

SUMMARY:
Impact of Maraviroc, a ART CCR5 inhibitor, on the intensification of immune function in HIV-1 infected subjects receiving immunisation with novel antigens

The purpose of the study is to investigate the impact of adding Maraviroc (an anti-HIV agent) to a participant's normal HIV medication, on immune function. As part of the study participants will also receive three different vaccinations and a skin test. The study will also look at whether Maraviroc influences the body's response to these.

The vaccines are given to stimulate the body's immune system, so we can therefore evaluate the impact that Maraviroc has on this.

The duration of the study will be just over 24 weeks plus a screening period up to 4 weeks prior to the start of the study.

DETAILED DESCRIPTION:
Maraviroc is a CCR5 antagonist with potent anti-HIV-1 activity, demonstrated in both treatment naïve and experienced settings. Binding of maraviroc to CCR5 leads to the loss of receptor function. Individuals with non-functioning CCR5 due to a 32 base pair deletion in the encoding gene are observed at a 1% frequency in the northern European Caucasian population. These individuals have near normal immune function, although differential response to renal transplant and West Nile virus have been reported relative to individuals with functional CCR5. The modest impact on immune function is indicative of a functional overlap between CCR5 and other CC chemokine receptors. While the precise role of CCR5 has not been established, data suggest a role in chemotaxis and inflammation.

An excess of clinical events, infective, inflammatory or malignant, have not been reported in persons receiving maraviroc relative to placebo or to efavirenz-based antiretroviral therapy over 48 weeks follow-up. Indeed, individuals randomized to maraviroc were noted in these studies to have modestly greater increases in CD4 T-cell numbers, not accounted for by changes in lymphocyte counts or rates of viral suppression.

The impact of inclusion of maraviroc in an antiretroviral treatment regimen on immune function has not been reported.

In chronically infected HIV-1+ individuals who progress to AIDS, the full functionality of the anti-HIV-1 CD8+ cytotoxic T lymphocyte response is progressively lost. This is accompanied by diminished responses to neo- and recall antigens and skin anergy (loss of DTH response). This is likely dependent on the loss of function and numbers of HIV-1-specific CD4+ helper T lymphocytes (Appay and Sauce 2008). This process is apparently, at least partially, irreversible despite otherwise successful, currently used antiretroviral drug regimens. Accumulation of functionally inert ('anergic') HIV-1-specific CD4+ and CD8+ CD28- CTLA-4hi T cells is observed, which lack proliferative and IL-2 producing ability and cytolytic function despite maintaining the capacity to produce IFN-γ (Deeks and Walker 2007). A balanced response in which the host responds appropriately to prevalent antigen, such as HIV-1 Gag, yet remains relatively quiescent, may prove to be the strongest functional correlate of virologic control (Imami et al. 2002; Imami et al. 2007).

Recent work has shown that tetanus antibody responses are significantly impaired in HIV patients on successful ART (Hart et al. 2007). A recently identified CD4 T-cell subset, known as follicular T cells (TFH) plays a crucial role in the development of humoral immune responses to protein antigens such as tetanus toxoid (King et al. 2008). Follicular CD4 T cells express a chemokine receptor called CXCR5, a protein called inducible co-stimulatory factor (ICOS) and are readily identified in peripheral blood. Follicular CD4 T cells are prone to activation induced cell death which is believed to be a major mechanism of CD4 T-cell depletion in chronic HIV-1 infection and therefore could be a vulnerable target in retroviral disease. A reduction in circulating CD4 TFH numbers and/or function may account for the failure of HIV-1 patients to respond to tetanus vaccination.

The aims of this study are to investigate the impact of the addition of maraviroc to a successful HIV-1 treatment regimen on in vitro (lymphoproliferative, ELISpot assays) and in vivo (response to subcutaneous and GI administered vaccination by antibody and skin tests as applicable) immune function, and to assess function of CD4 TFH cells by measuring cytokine and co-stimulatory protein expression in this T-cell subset.

This 92 patient randomized, blinded placebo controlled trial plans to investigate the impact of the addition of maraviroc to on-going successful PI/r based ART, with regards to multiple immunology markers including markers of activation, CD4 and CD8 T-cell subsets, immune function (Elispot and lymphoproliferative responses to HIV-1 and recall antigens and/or peptides (Gag, TTox, CMV), and antibody response to oral (cholera) and deep subcutaneous/IM (meningococcus) neoantigens and recall antigens (Tetanus toxoid)) and to assess function of CD4 TFH cells by measuring cytokine and co-stimulatory protein expression in this subset. Delayed type hypersensitivity will be tested at baseline and week 24, and read 48 hours post administration of the Mantoux test.

Participants will be stratified by CD4 nadir, with 50% of patients having a CD4 nadir <200 cells/µl blood.

Maraviroc will be administered to patients at a dose level of 150mg BID. This dose is approved for use in the UK.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 antibody positive
* On a virologically suppressive regimen for at least 24 weeks and stable on a PI/r (ATV, LPV or DRV) plus Truvada or Kivexa for at least 4 weeks prior to screening
* Current HIV-1 RNA <50cps/ml plasma on 2 occasions >4 weeks apart
* No prior CCR5 or CXCR4 antagonist use
* Prior tetanus toxoid immunisation or known tetanus antibodies. Immunisation must have taken place in the past 10 years, but not within 1 month of baseline visit.
* Known CD4 nadir
* If the subject is a woman of child bearing potential, she must agree to use a double barrier method of contraception
* Willing and able to provide written informed consent
* At least 18 years old

Exclusion Criteria:

* Current or prior immunologically active agents (use of IL-2, GH or GHRH, corticosteroids (except inhaled), G- and GM-CSF) deemed to potentially impact study results.
* History of HIV, cholera or meningococcal immunisation
* Other known immune deficiency or use of immune suppressant
* History of malignancy (except low volume Kaposi's sarcoma) or chemotherapy
* Contraindication to maraviroc
* Peanut or soya allergy
* Antiretroviral agents other than those in inclusion list
* Drugs known to reduce exposure to maraviroc (CYP3A inducers)
* Contraindication to vaccines or vaccine components and/or components of skin test kits
* Pregnant or lactating or planning to become pregnant during the study period
* Acute feverish, stomach or intestinal illness
* Received an investigational medicinal product as part of a clinical trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes in tetanus antibody titres following vaccination | 24 weeks

SECONDARY OUTCOMES:
Changes in composite lymphocyte proliferation responses by group | 24 weeks
CD4 and CD8 subsets, activation and co-stimulation markers, plasma RNA viral load (pVL) | 24 weeks
Response to oral and subcutaneous neoantigens and recall antigens | 24 weeks
Influence on CCR5 antagonism on CD4 follicular T-cell counts and function | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Moyle, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom